CLINICAL TRIAL: NCT02478411
Title: Functional and Motor Effects of an Early Cycloergometric Physiotherapy Program in Critically Ill Patients With Invasive Mechanical Ventilation. A Randomized Controlled Trial
Brief Title: Early Cycloergometric Physiotherapy in Critically Ill Patients With Invasive Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Son Llatzer (Other)
Responsible Party: Principal Investigator, Gemma Rialp, M.D., Hospital Son Llatzer
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CYCLE-ICU-001
Record Dates: First submitted 2015-06-14; First posted 2015-06-23 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Weakness
Keywords: muscle weakness; rehabilitation; intensive care; mechanical ventilation; cyclo ergometer; physiotherapy
MeSH Terms: conditions — Asthenia; Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cycle ergometer physiotherapy (Experimental): 15 minutes of cycle ergometer physiotherapy plus 15 minutes of conventional physiotherapy, once daily, five days a week, as long as patients remain in the intensive care unit
  Interventions: Procedure: Cycle ergometer physiotherapy
- Conventional physiotherapy (Active Comparator): 30 minutes of conventional physiotherapy, once daily, five days a week, as long as patients remain in the intensive care unit
  Interventions: Procedure: Conventional physiotherapy

INTERVENTIONS:
Procedure: Cycle ergometer physiotherapy — 15 minutes of cyclo ergometer physiotherapy with MOTOmed ® Letto 2 device with passive, motor-assisted and active-resisted exercise of the lower and upper extremity, and 15 minutes of conventional physiotherapy
  Other Names: MOTOmed ® Letto 2
  Arms: Cycle ergometer physiotherapy
Procedure: Conventional physiotherapy — 30 minutes of conventional physiotherapy
  Arms: Conventional physiotherapy

SUMMARY:
Study designed to evaluate the functional and motor effects in critically ill subjects at ICU and hospital discharge with the incorporation of a mobilization program of cycloergometric physiotherapy sessions compared with conventional physiotherapy.

DETAILED DESCRIPTION:
Cycloergometric treatment is described to improve the functional and motor status of critically ill subjects. However, there are few studies comparing cycloergometric physiotherapy and conventional physiotherapy in intensive care subjects under mechanical ventilation. The most relevant of these studies conducted by Burtin et al showed beneficial effects of cycloergometric treatment. However, the duration of the physiotherapy sessions in this study differed between groups as cycloergometric group received a double daily dose of treatment. It is known that the intensity of physiotherapy also affects the functional and motor status.

For this reason, the investigators designed a randomized controlled study with early cycloergometric or conventional treatment, with the same intensity between groups to analyze objective functional and motor endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Criteria of functional independence before hospital admission (Barthel scale > 70 points).
* Invasive mechanical ventilation < 72 hours.
* Signed informed consent.

Exclusion Criteria:

* Neuromuscular disease (peripheric or central neurologic disorder).
* Presumed fatal evolution in 48 hours.
* Conditions that impede pedaling movement (leg, pelvis or lumbar spinal surgery or traumatism).
* Admission due to cardiac arrest.
* Pregnancy.
* Thrombopenia less than 50.000.
* Severe agitation.
* Hemodynamic instability with noradrenaline requirements greater than 1 mcg/kg/min.
* Fraction of inspired Oxygen (FiO2) requirements greater that 0.55 and respiratory rate greater than 30 bpm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2015-06; Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Walking test distance at six minutes | At hospital discharge, with an expected average of 4 weeks after hospital admission
Short Form-36 Health Survey (SF-36), physical functioning section | At 28 days after hospital discharge, that is an expected average of 8 weeks
Basic activities of daily living score (BADL) | At 28 days after hospital discharge, that is an expected average of 8 weeks

SECONDARY OUTCOMES:
Lung Functional Testing | At the end of hospital stay, with an expected average of 5 weeks
Presence of intensive care acquired paresis (Medical Research Council score < 48 points) | During ICU admission and ICU discharge, with an expected average of 2 weeks
ICU mobilization scale | During hospital stay, as expected average of 4 weeks, and at 28 days and at 6 months after discharge
Isometric quadriceps force (N/kg) | During ICU admission, with an expected average of 2 weeks
  Quadriceps strength will be measured with a handheld dynamometer with patients in supine position and 30º of knee flexion.
Walking test distance at six minutes | At 28 days and at 6 months after hospital discharge, that is up to 1 year
Short Form-36 Health Survey (SF-36), physical functioning section | At 7 days and at 6 months after hospital discharge, that is up to 1 year
Basic activities of daily living score (BADL) | At 7 days and at 6 months after hospital discharge, that is up to 1 year

OTHER OUTCOMES:
Changes in Pulse Oximeter Oxygen Saturation (SpO2) between end and initial values after physiotherapy sessions | ICU admission, with an expected average of 2 weeks
Change in respiratory rate between end and initial values after physiotherapy sessions | ICU admission, with an expected average of 2 weeks
  Respiratory rate
Change in heart rate between end and initial values after physiotherapy sessions | ICU admission, with an expected average of 2 weeks
Change in mean blood pressure between end and initial values after physiotherapy sessions | ICU admission, with an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Rialp, M.D., Principal Investigator — IDISPA
Locations (1):
- Hospital Son llàtzer, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Result] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Result] TEAM Study Investigators; Hodgson C, Bellomo R, Berney S, Bailey M, Buhr H, Denehy L, Harrold M, Higgins A, Presneill J, Saxena M, Skinner E, Young P, Webb S. Early mobilization and recovery in mechanically ventilated patients in the ICU: a bi-national, multi-centre, prospective cohort study. Crit Care. 2015 Feb 26;19(1):81. doi: 10.1186/s13054-015-0765-4. PMID 25715872
- [Result] Schweickert WD, Kress JP. Implementing early mobilization interventions in mechanically ventilated patients in the ICU. Chest. 2011 Dec;140(6):1612-1617. doi: 10.1378/chest.10-2829. PMID 22147819
- [Result] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Result] Needham DM, Truong AD, Fan E. Technology to enhance physical rehabilitation of critically ill patients. Crit Care Med. 2009 Oct;37(10 Suppl):S436-41. doi: 10.1097/CCM.0b013e3181b6fa29. PMID 20046132
- [Result] Burtin C, Clerckx B, Robbeets C, Ferdinande P, Langer D, Troosters T, Hermans G, Decramer M, Gosselink R. Early exercise in critically ill patients enhances short-term functional recovery. Crit Care Med. 2009 Sep;37(9):2499-505. doi: 10.1097/CCM.0b013e3181a38937. PMID 19623052
- [Result] Bourdin G, Barbier J, Burle JF, Durante G, Passant S, Vincent B, Badet M, Bayle F, Richard JC, Guerin C. The feasibility of early physical activity in intensive care unit patients: a prospective observational one-center study. Respir Care. 2010 Apr;55(4):400-7. PMID 20406506